CLINICAL TRIAL: NCT03842748
Title: Non-invasive Diagnostic Model of Liver Fibrosis Associated With Non-alcoholic Fatty Liver Disease and Prediction of Prognosis
Brief Title: Non-invasive Diagnostic Model of Liver Fibrosis Associated With NAFLD and Prediction of Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, Minghui Li, Head of Liver Diseases Center, Beijing Ditan Hospital
Other Study IDs: XXZ0302
Record Dates: First submitted 2019-01-19; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Nonalcoholic; fatty liver; hepatitis; liver fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Hepatitis; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 192 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective study group: 200 patients with non-alcoholic fatty liver disease, fatty liver hepatitis, and fibrosis have been identified for pathological diagnosis of liver histology and without other liver diseases. Before liver biopsy were performed, liver function, coagulation function, renal function, blood glucose, blood lipids, liver elasticity measurement, imaging indicators and demographic data were detected and recorded. To evaluate diagnostic ability of current non-invasive diagnostic model of NAFLD fibrosis and adaptability of model indicators to diagnosis of these patients, and correct the indicators including discarding unsuitable and incorporating new indicators and adjusting the diagnostic score. Establish a non-invasive diagnostic model for liver fibrosis in Beijing based on NAFLD.
- Prospective observational study group: 100 patients without other liver diseases and ultrasound-tested fatty liver were enrolled, and histopathological diagnosis of liver were included , and liver function, coagulation function, renal function, blood glucose, and non-invasive model analysis, blood lipids, liver elasticity measurements and imaging indicators were examined and demographic data were collected. Adjusted the index of non-invasive diagnostic model to further revise and improve the diagnostic efficacy of diagnostic model. Long-term follow-up observations were performed in the prospective observation cohort. To explore the correlation and predictive ability of noninvasive diagnostic models for long-term outcomes of disease. Finally, a model for predicting the outcome of progression of liver fibrosis in NAFLD was established.

SUMMARY:
In a retrospective study, 200 patients with non-alcoholic fatty liver disease, fatty liver hepatitis, and fatty liver fibrosis have been identified for pathological diagnosis of liver histology and exclusion of other liver diseases. Before the liver biopsy were performed, these patients should detect liver function, coagulation function, renal function, blood glucose, blood lipids, liver elasticity measurement and imaging indicators and results, and demographic data. To evaluate the diagnostic ability of the current non-invasive diagnostic model of NAFLD fibrosis and the adaptability of model indicators to the diagnosis of enrolled patients, and to correct the indicators, including discarding unsuitable indicators and incorporating new indicators, and adjusting the diagnostic score. Establish a non-invasive diagnostic model for liver fibrosis in Beijing based on NAFLD. In a prospective observational study, 100 patients without other liver diseases and ultrasound-tested fatty liver were enrolled, and histopathological diagnosis of liver were included in the study, and liver function, coagulation function, renal function, blood glucose, and non-invasive model analysis were detected. Blood lipids, liver elasticity measurements, and imaging indicators were examined and demographic data were collected. The non-invasive diagnostic model established by retrospective study was used to diagnose fibrosis and its staging, compared with histopathological diagnosis, and adjusted the index of non-invasive diagnostic model to further revise and improve the diagnostic efficacy of the diagnostic model. Long-term follow-up observations were performed in the prospective observation cohort. The liver function, coagulation function, renal function, blood glucose, blood lipids, liver elasticity and imaging examination were performed during the observation period, and the treatment events and the progress of the patients were recorded. To explore the correlation and predictive ability of noninvasive diagnostic models for long-term outcomes of disease. Finally, a model for predicting the outcome of progression of liver fibrosis in NAFLD was established.

DETAILED DESCRIPTION:
This topic is a prospective - retrospective observational study including two parts, retrospective and prospective: in a retrospective study, 200 patients with non-alcoholic fatty liver disease, fatty liver hepatitis, and fatty liver fibrosis have been identified for pathological diagnosis of liver histology and exclusion of other liver diseases. The liver biopsy performed in the enrolled patients included liver function, coagulation function, renal function, blood glucose, blood lipids, liver elasticity measurement and imaging indicators and results, and demographic data. To evaluate the diagnostic ability of the current non-invasive diagnostic model of NAFLD fibrosis and the adaptability of model indicators to the diagnosis of enrolled patients, and to correct the indicators, including discarding unsuitable indicators and incorporating new indicators, and adjusting the diagnostic score. Establish a non-invasive diagnostic model for liver fibrosis in Beijing based on NAFLD. In a prospective observational study, 100 patients without other liver diseases and ultrasound-tested fatty liver were enrolled, and histopathological diagnosis of liver were included in the study, and liver function, coagulation function, renal function, blood glucose, and non-invasive model analysis were included. Blood lipids, liver elasticity measurements, and imaging indicators were examined and demographic data were collected. The non-invasive diagnostic model established by retrospective study was used to diagnose fibrosis and its staging, compared with histopathological diagnosis, and adjusted the index of non-invasive diagnostic model to further improve and improve the diagnostic efficacy of the diagnostic model. Long-term follow-up observations were performed on the prospective observation cohort. The liver function, coagulation function, renal function, blood glucose, blood lipids, liver elasticity and imaging examination were performed during the observation period, and the treatment events and the progress of the patients were recorded. To explore the correlation and predictive ability of noninvasive diagnostic models for long-term outcomes of disease. Finally, a model for predicting the outcome of progression of liver fibrosis in NAFLD was established.

ELIGIBILITY:
Inclusion Criteria:

1. patients with non-alcoholic fatty liver, fatty liver hepatitis and fatty liver fibrosis: all meet the diagnostic criteria of China's "Guidelines for the Prevention and Treatment of Non-alcoholic Fatty Liver Diseases (2018 Update)";
2. Age between 18 and over 75;
3. patient were never treated with no hormones and / or immunosuppressants and other liver protection drugs.

Exclusion Criteria:

1. combined with hepatitis virus infection;
2. autoimmune liver disease;
3. HIV infection;
4. long-term alcohol abuse and / or other liver damage drugs;
5. mental illness;
6. Evidence of liver tumors (liver cancer or AFP > 100 ng/ml);
7. decompensated cirrhosis;
8. Serious diseases such as heart, brain, lung, kidney, etc. can not participate in long-term follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject of this study was patients with non-alcoholic fatty liver, fatty liver hepatitis and fatty liver fibrosis diagnosed by histopathology of the liver. Patients enrolled in the study excluded other liver diseases such as alcoholic fatty liver and hepatitis, viral hepatitis. , autoimmune diseases, drug-induced hepatitis and liver cancer.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between clinical biochemical parameters of nonalcoholic fatty liver disease and pathological diagnosis of liver perforation | at baseline, 24weeks, 48weeks, 72weeks, 96weeks, 120weeks, 144weeks, 168weeks, 192weeks.
  Correlation between clinical biochemical parameters of nonalcoholic fatty liver disease and pathological diagnosis of liver perforation, and the change of clinical biochemical parameters of nonalcoholic fatty liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Li, master, Principal Investigator — Liver Diseases Center, Beijing Ditan Hospital, Capital Medical University
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality, China